CLINICAL TRIAL: NCT04352296
Title: Effect of Individualized Versus Standard Blood Pressure Management During Mechanical Thrombectomy for Anterior Ischemic Stroke
Brief Title: Effect of Individualized Versus Standard Bp Management During MT for Anterior Ischemic Stroke
Acronym: DETERMINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BMR_2020_12
Record Dates: First submitted 2020-04-10; First posted 2020-04-20 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Acute Cerebrovascular Accident
Keywords: Acute ischemic stroke; Large vessel occlusion; Mechanical thrombectomy; Blood pressure management; Brain infarction; Endovascular procedure; Thrombectomy; Blood pressure; Low blood pressure; Hemodynamic; Hypertension
MeSH Terms: conditions — Stroke; Ischemic Stroke; Brain Infarction; Hypotension; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Individualized BP management during mechanical thrombectomy with the administration of diluted norepinephrine (5-10 µg/ml) or nicardipine (1 mg/ml) or urpidil (5 mg/ml) to maintain the MAP within 10% of the first MAP measured in the angiography suit.
  Interventions: Procedure: Individualized blood pressure
- Control group (Active Comparator): Standard BP management based on international guidelines: Treatment of hypotension defined by a systolic blood pressure <140 mm Hg, and treatment of hypertension defined by a systolic blood pressure > 180 mm Hg or diastolic blood pressure >105 mm Hg) with usual treatments (norepinephrine, ephedrine or phenylephrine for hypotension; intravenous nicardipine or uradipil for hypertension).
  Interventions: Procedure: Standard blood pressure

INTERVENTIONS:
Procedure: Individualized blood pressure — Individualized blood pressure management during mechanical thrombectomy with the administration of diluted norepinephrine (5-10 µg/ml) or nicardipine (1 mg/ml) or urpidil (5 mg/ml) to maintain the MAP within 10% of the first MAP measured in the angiography suit
  Arms: Experimental group
Procedure: Standard blood pressure — Standard blood pressure management based on international guidelines: Treatment of hypotension defined by a systolic blood pressure <140 mm Hg, and treatment of hypertension defined by a systolic blood pressure > 180 mm Hg or diastolic blood pressure >105 mm Hg) with usual treatments (norepinephrine, ephedrine or phenylephrine for hypotension; intravenous nicardipine or uradipil for hypertension).
  Arms: Control group

SUMMARY:
DETERMINE is a multicenter, prospective, randomised, open, blinded end-point assessed (PROBE) trial, to evaluate two approaches of blood pressure (BP) management during mechanical thrombectomy for acute ischemic stroke due to an anterior large vessel occlusion.

DETAILED DESCRIPTION:
This study have to objective to evaluate the efficacy of an individualized BP control during mechanical thrombectomy (regardless of the sedation modality), by maintaining a mean arterial pressure (MAP) within 10% of the first MAP measured in the angiography suit, compared to the standard BP management, on the 3-month functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Acute ischemic stroke due to an anterior large vessel occlusion: occlusion of the M1 or M2 segments of the middle cerebral artery, anterior cerebral artery (A1 segment), intracranial internal carotid artery, or tandem occlusions.
* Indication for mechanical thrombectomy under general anesthesia or conscious sedation within the first 6 hours from symptoms onset or within the first 24 hours if DAWN or DEFUSE-3 criteria are met.
* Affiliation to social security assurance.

Exclusion Criteria:

* Contre-indication to mechanical thrombectomy
* Intubation or induction of general anaesthesia prior to randomization
* Acute ischemic strokes associated with a posterior circulation large vessel occlusion (basilar artery, vertebral artery, posterior cerebral artery)
* Intra-hospital onset of acute ischemic stroke, or secondary to a medical, interventional or surgical procedure (interventional cardiology, cardiac or vascular surgery) or any post-surgery ischemic stroke.
* Pre-existing neurological disability limiting neurological assessment at 3 months: mRS >2 at randomization.
* Contraindication to iodinated contrast agents
* Known pregnancy or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — woman and man
Enrollment: 433 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Number of patient with a favorable functional outcome at 3 months | 3 months visit
  Rankin score less than 3

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Dr Maier, Principal Investigator — Hopital Fondation A de Rothschild; Etienne Dr Gayat, Study Chair — Hôpital Lariboisière, AP-HP; Morgan Dr Leguen, Study Chair — Hôpital Foch; Russel Dr Chabanne, Study Chair — CHU Gabriel Montpied; Baptiste Dr Balanca, Study Chair — Hospices Civils de Lyon, Hôpital Pierre Wertheimer; Benoit Pr Tavernier, Study Chair — Hôpital Roger Salengro, Lille; Thomas Pr Geeraerts, Study Chair — Hôpital Purpan, CHU Toulouse; Benjamin Pr Gory, Study Chair — "Centre Hospitalier Régional Universitaire (Nancy); Grégoire Dr Boulouis, Study Chair — Centre Hospitalier Régional Universitaire de Tours; Vincent Pr Degos, Study Chair — La Pitié Salpêtrière (APHP); Gaultier Dr Marnat, Study Chair — CHU de Bordeaux, Hôpital Pellegrin
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maier B, Gory B, Chabanne R, Tavernier B, Balanca B, Audibert G, Thion LA, Le Guen M, Geeraerts T, Calviere L, Degos V, Lapergue B, Richard S, Djarallah A, Mophawe O, Boursin P, Le Cossec C, Blanc R, Piotin M, Mazighi M, Gayat E; DETERMINE Investigators. Effect of an individualized versus standard blood pressure management during mechanical thrombectomy for anterior ischemic stroke: the DETERMINE randomized controlled trial. Trials. 2022 Jul 26;23(1):598. doi: 10.1186/s13063-022-06538-9. PMID 35883180